CLINICAL TRIAL: NCT06782217
Title: Prospective Observational Study to Evaluate the Safety of Immunotherapy as a Treatment for Hymenoptera Venom Allergy
Status: Recruiting | Type: Observational
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Other Study IDs: ITK-VENOX-2024-01
Record Dates: First submitted 2024-09-16; First posted 2025-01-17 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Allergy, Insect Venom; Allergy Insect Stinging; Insect Sting Allergy
Keywords: Allergy; Immunothepary; Apis mellifera; Vespula spp.; Insect venom
MeSH Terms: conditions — Venom Hypersensitivity; Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum to perform immunological study of total IgE, and specific IgE, IgG4, IgG1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients allergic to hymenoptera venom: Patients allergic to hymenoptera venom and receive the clinical recommendation to be treated with VENOX immunotherapy (ATC code: V01AA07).
  Interventions: Biological: VENOX

INTERVENTIONS:
Biological: VENOX — Treatment with allergy vaccine againts Vespula spp. (wasp) or Apis mellifera (bee), as per clinical indication.

SUMMARY:
Observational study to evaluate the safety of immunotherapy as a treatment for Hymenoptera venom allergy, analyzing the adverse reaction to immunotherapy as well as the allergic reaction to a spontaneous hymenoptera sting. This study will be conducted in Spain (multicentric) and data will be collected prospectively.

DETAILED DESCRIPTION:
Observational study to evaluate the adverse reaction to immunotherapy as well as the allergic reaction to a spontaneous hymenoptera sting (safety evaluation), also it will be evulated the quality of life of the patient using one QoL questionnair before and after immunotherapy treatment.

The patients aged equal or more than 14 years old, not gender differentiation, and sensitised to heminoptera venom. The total number of participants is expected to be 120.

This study will be conducted in Spain (multicentric) and data will be collected prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. The study population consisted of allergic participants indicated for treatment with immunotherapy with hymenoptera venom (Apis mellifera or Vespula spp.) according to standard clinical practice.
2. Age equal to or older than 14 years, without gender differences.
3. Not having received immunotherapy with hymenoptera venom in the previous 5 years.
4. That they agree to participate in the study and sign the informed consent form. In the case of minors, the parent or guardian of the participant must also sign the informed consent form.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Having received immunotherapy with hymenoptera venom during the 5 years prior to the start of the study.
3. Participants who do not agree to participate and/or do not sign the informed consent form.
4. Participants who do not comply with the medical indications or do not show cooperation with respect to the immunotherapy treatment.
5. Participants with oncological diseases under active treatment or with autoimmune diseases under immunosuppressive treatment.
6. Participants in whom the administration of immunotherapy is contraindicated.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants aged 14 years and older diagnosed with allergy to Apis mellifera and/or Vespula spp. venom, susceptible to receive immunotherapy wit himenoptera venom according to standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-Emergent adverse reactions (safety and tolerability) in patients diagnosed with allergy to hymenoptera venom (Apis mellifera and/or Vespula spp.) with indication to receive immunotherapy with the causative venom. | 12 months
  Evaluation of the severity of reactions in relation to subcutaneous immunotherapy following the indications proposed by the World Allergy Organization (WAO).

SECONDARY OUTCOMES:
Evaluation of the immunogenicity of the participant after 6 and 12 months of treatment. | 12 months
  Immunological study: total IgE, and specific IgE, IgG4, IgG1 (total extract and molecular components of Vespula spp. and Apis mellifera). The immunological analysis will be performed according to the usual clinical practice of the center and the serum samples will be stored for the complete analysis in the facilities of the sponsor, using the ALEX technique.
Quality of life in treated participants after 6 and 12 months of treatment. | 12 months
  Questionnaire of "Quality of Life in People Allergic to Hymenoptera Venom" (HiCaVi), property/copyright of SEAIC (Sociedad Española de Alergología e Inmunología Clínica).
  The quality of life questionnaire consists of 14 questions, the first nine questions are mandatory. The score for each question is inverse to the order of the answer, i.e., the first answer scores 7 and the seventh answer scores 1.
  The score shall be obtained by adding up all the questions answered and dividing by the total number of questions answered.
  The total score goes from 1 to 7, being the 1 the worst quality and the 7 the best one.
Evaluation of the effectiveness of treatment with immunotherapy, once the maintenance dose of 100 μg/mL is reached, in participants suffering spontaneous natural repicures during the 1-year follow-up. | 12 months
  Registration of allergic reactions after spontaneous natural stings.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Javier Carballada, MD, Principal Investigator — Hospital Universitario Lucus Augusti
Locations (9):
- Spain (9):
  - Hospital Arquitecto Marcide, Ferrol, A Coruña
  - Hospital Virgen del Puerto Plasencia, Plasencia, Cáceres
  - Hospital Público Da Mariña, Burela de Cabo, Lugo
  - Hospital Comarcal de Monforte de Lemos, Monforte de Lemos, Lugo
  - Hospital de A Coruña, A Coruña
  - Hospital Vall d' Hebron, Barcelona
  - Hospital Universitario Lucus Augusti, Lugo
  - Complejo Hospitalario Universitario de Ourense, Ourense
  - Hospital Universitario de Pontevedra, Pontevedra

REFERENCES:
- [Background] Oude Elberink JN, De Monchy JG, Van Der Heide S, Guyatt GH, Dubois AE. Venom immunotherapy improves health-related quality of life in patients allergic to yellow jacket venom. J Allergy Clin Immunol. 2002 Jul;110(1):174-82. doi: 10.1067/mai.2002.125827. PMID 12110838
- [Background] Golden DB. Insect sting allergy and venom immunotherapy: a model and a mystery. J Allergy Clin Immunol. 2005 Mar;115(3):439-47; quiz 448. doi: 10.1016/j.jaci.2005.01.005. PMID 15753884
- [Background] Bousquet J, Muller UR, Dreborg S, Jarisch R, Malling HJ, Mosbech H, Urbanek R, Youlten L. Immunotherapy with Hymenoptera venoms. Position paper of the Working Group on Immunotherapy of the European Academy of Allergy and Clinical Immunology. Allergy. 1987 Aug;42(6):401-13. doi: 10.1111/j.1398-9995.1987.tb00355.x. PMID 3310714
- [Background] Demsar Luzar A, Korosec P, Kosnik M, Zidarn M, Rijavec M. Hymenoptera Venom Immunotherapy: Immune Mechanisms of Induced Protection and Tolerance. Cells. 2021 Jun 22;10(7):1575. doi: 10.3390/cells10071575. PMID 34206562